CLINICAL TRIAL: NCT06778122
Title: A Series of N-of-1 Randomised, Adaptive, Blinded, Placebo-Controlled Trials of Overnight In-Bedroom Air Filtration as Adjuvant Treatment in Reducing Inflammatory Biomarkers Among Survivors of Adult-Onset Cancer With Elevated C-Reactive Protein
Brief Title: In-Bedroom Renewed Air as Anti-inflammatory Adjuvant Therapy in Cancer Survivors
Acronym: BREATHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: IQAir AG (Unknown); PremaLabs Diagnostics, Ltd (Unknown); A&D Instruments, Ltd (Unknown); Lansion Biotechnology Co. Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 22105/001
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-01

CONDITIONS: Cancer Survivors; Cardiotoxicity; Cardiovascular Toxicity Induced by Antitumoral Drugs
Keywords: Cancer survivors; Cardio-oncology rehabilitation; Inflammation; Air filtration systems; Air purifiers
MeSH Terms: conditions — Cardiotoxicity; Inflammation

STUDY DESIGN:
Intervention Model Description: N-of-1 trial design (multiple crossover trial design for single participants). N-of-1 series (aggregated N-of-1 trial). Each participant will be randomly allocated to 3 treatment sets or cycles, each comprising a 14-day period of active therapy and a 14-day period of sham intervention (placebo - standard of care).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The sequence allocation will be masked for the participants, general practitioners, primary care staff and research team members, except for the field researcher to dispense the correct treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Air purifier nightly (Active Comparator): Participants are exposed to filtered air (HyperHEPA filter) nightly in the bedroom, in 14-day periods, up to 3 treatment sets in 12 weeks (blinded phase).
  The blinded N-of-1 trial will last between 4 and 12 weeks per participant, depending on the treatment set(s) received (cycle 1, 2 and 3) to produce evidence of clinical benefit (CRP < 2 mg/L or CRP reductions ≥ 35%).
  Interventions: Device: High efficiency particulate air filtration system (nightly administration)
- Sham air filter (Sham Comparator): Participants receive an intervention of sham air purifiers nightly in the bedroom, in 14-day periods, up to 3 treatment sets in 12 weeks (blinded phase). The blinded N-of-1 trial will last between 4 and 12 weeks per participant, depending on the treatment set(s) received (cycle 1, 2 and 3) to produce evidence of clinical benefit (CRP < 2 mg/L or CRP reductions ≥ 35%).
  Interventions: Device: Air filtration system without filters (sham)
- Air purifier nightly and daily (Experimental): Participants are exposed to nightly and daily filtered air (HyperHEPA filter) in the bedrooms (open-label phase). The air purifier with active filter is continuously operated (24 hours for 14 days). Participants who do not achieve the clinically meaningful change established in the trial (CRP < 2 mg/L or CRP reductions ≥ 35%) after the treatment set 3 (cycle 3) will take this open-label phase.
  Interventions: Device: High efficiency particulate air filtration system (nightly and daily administration)
- No treatment (No Intervention): 14-day period of no intervention. Participants who do not achieve the clinically meaningful change established in the trial (CRP < 2 mg/L or CRP reductions ≥ 35%) after the treatment set 3 (cycle 3) will take this open-label phase.

INTERVENTIONS:
Device: High efficiency particulate air filtration system (nightly administration) — Portable air purifier is programmed to provide a dose of filtered air at 275 m³/h nightly for at least 7 hours consecutive within a time window between 10:00 p.m. and 10:00 a.m. Air purifier is set up with active filters (HyperHEPA technology). Dose adjustments are permitted in the study where noise disturbance is an issue for participants. The air filtration therapy will be delivered in doses decreasing sequentially in terms of speed mode. Participants will be instructed to keep doors and windows of the bedroom closed during each session at night, and to follow a similar bedtime routine.
  Arms: Air purifier nightly
Device: High efficiency particulate air filtration system (nightly and daily administration) — Portable air purifier set up with active filters (HyperHEPA technology) is continuously in operation (24 hours for 14 days) at 275 m³/h in bedrooms with the door and windows closed. During this open-labell phase, the participants will be asked to remain in the bedroom for as long as possible and to keep an activity log for the outdoor locations. Dose adjustments are permitted.
  Arms: Air purifier nightly and daily
Device: Air filtration system without filters (sham) — Portable air purifier is programmed to provide a dose of filtered air at 275 m³/h nightly for at least 7 hours consecutive within a time window between 10:00 p.m. and 10:00 a.m. Air purifier is set up with a sham filter, which is identical in appearance and noise as the HyperHEPA filter (active filter) when the air purifier is in operation. Dose adjustments are permitted in the study where noise disturbance is an issue for participants.
  Arms: Sham air filter

SUMMARY:
The BREATHS trial aims to investigate whether overnight in-bedroom air filtration reduces inflammation and cardiac biomarkers in adult survivors of cancer who are at high risk for cardiovascular complications.

The study consists of individualized experiments (N-of-1 trials) conducted in the home settings of adults residing in densely populated urban areas with the most severe air quality levels in Valencia, Spain, where fine particulate matter (PM2.5) and nitrogen dioxide levels exceed the limits set by the World Health Organization (WHO) and EU Directive.

Participants will be exposed to 3 treatment sets (blinded phase), each consisting of a 14-day period of filtered air using a portable air filtration unit ("true-HyperHepa) and a 14-day period of unfiltered air (using the same portable unit with "sham filters"). The intervention will be administered nightly for a minimum of 7 consecutive hours and will last between 4 and 12 weeks for each participant, contingent upon the demonstration of clinical benefit, defined by a reduction in the levels of the blood biomarker C-reactive protein. An unblinded phase will be implemented for participants who do not experience a clinically meaningful change in CRP. During this phase, they will undergo a 14-day period without treatment, followed by 14-day period of both nightly and daily filtered air therapy.

The primary endpoint of this study is defined as the change in blood concentrations of CRP. The secondary endpoints include the changes in levels of three other noninvasive blood biomarkers associated with inflammation and cardiovascular health, and blood pressure.

Both indoor and outdoor fine particulate matter (PM2.5) exposure concentrations will be continuously monitored in the study.

DETAILED DESCRIPTION:
Background. Inflammation, a common result of anticancer therapies, correlates with poor survival and cardiovascular issues in cancer survivors. High levels of C-reactive protein (CRP), D-dimer, and serum amyloid A (SAA) indicate cancer recurrence, mortality, and cardiotoxicity. CRP-lowering clinical trials have proven that the magnitude of the reduction in cardiac events in patients with residual inflammatory risk is directly proportional to the achieved reduction in CRP, with the greatest benefit in those achieving a threshold below than 2 milligrams per litre (mg/L).

Cancer survivors may benefit from non-pharmacological anti-inflammatory treatments that do not exacerbate cardiotoxicity burden. Evidence suggests the air purifiers lower inflammatory biomarkers in high-risk cardiovascular groups. Air filtration presents a promising alternative to inflammation-inhibiting drugs, but its anti-inflammatory and cardioprotective effects in cancer survivors and interactions with medications remain unclear.

Design, setting and participants. A series of N-of-1 randomised, adaptive, blinded, placebo-controlled trials will be conducted at the home sitting of community-dwelling cancer survivors who are registered in primary care practices of the city of Valencia, Spain. Participants eligible are aged 18 years or older, have a history of breast, colorectal, prostate, lung and haematologic cancer, completed curative cancer treatment with evidence of remission and screened blood CRP level of at least 3 mg/L (within individual SD CRP of ~0.20 mg/L at baseline is accepted).

Screening for CRP levels. Up to two home visits could be carried out to collect a 5 microlitres (µl) blood microsample and analyse the CRP levels in real-time of the potentially eligible participants. These screening visits will be done no more than 28 and 7 days prior to blinded N-of-1 phase, respectively.

Recruitment. Participants will be identified via 3 strategies: advertisements on social media, snowball sampling and in-primary care clinics referrals. Staff from local primary care setting participating in the study will identify eligible potentially participant. The selection criteria for primary care settings were based on neighborhood air quality, specifically urban areas with the highest index impact of pollutant on population > 125 and NO2 levels exceeding WHO and EU Directive 2008/50/EC limits: Malilla, Russafa, and Arrancapins.

Intervention. Each participant will be randomly allocated (1:1 ratio per cycle) to 3 treatment sets, each comprising a 14-day period of active therapy (portable air filtration unit [PAFU] at 275 m3/h) and a 14-day period of placebo (unit with sham filters - standard of care) in the bedroom. Active therapy and placebo will be nightly administered during at least 7-hours consecutive within a time window between 10:00 p.m. and 10:00 a.m. The blinded N-of-1 trial enrolment will be between 4 and 12 weeks per participant, depending on the treatment set(s) received to produce evidence of clinical benefit (CRP < 2 mg/L or CRP reductions ≥ 35%) .

After 2-weeks wash-out period of the last blinded treatment set, participants who do not achieve a clinically meaningful change will be given an open-label phase to take 14-days of no treatment and 14-days of nightly and daily active therapy - the PAFU will be continuously operated (filtered air at 275 m3/h) in bedrooms with the door and windows closed. The nightly active therapy keeps the same as the blinded treatment sets and participants will be asked to remain in the bedrooms for as long as possible (e.g., nap time). Time exposed to the in-bedroom air quality will be recorded.

Outcomes measures. The primary outcome is the level change in CRP after air filtration treatment compared with placebo. The secondary outcomes are changes in D-dimer, SAA and HbA1c concentrations, and systolic and diastolic BP. Primary and secondary outcomes will be collected at baseline and in the day 7 and 14 of each period using at-home minimally invasive medical devices.

Self-reported questionnaires. Four short versions of self-reported questionnaires will be weekly completed as potential inflammation modifying confounding factors: Godin Leisure-Time Exercise Questionnaire (GLTEQ), Food Frequency Questionnaire (FFQ), Pittsburg Sleep Quality Index (PSQI) and in-home Patterns & Time-Activity Questionnaire (PTAQ).

In-bedroom and outdoor air quality measurement. The changes in airborne pollutants will be continuously measured in real-time throughout the trial period using two monitors that integrates a combination of sensors, including particulate matter.

Statistical plan. Following treatment set 1 and 2, interim analysis will be conducted to establish whether the active treatment, as compared with placebo, is clinically effective: achievement of CRP levels < 2 mg/L or CRP reductions ≥ 35%. While participants who achieve this clinically meaningful change will be discontinued of the N-of-1 trial, those who do not achieve it in the treatment set 3 will be given the open-label phase.

Changes from baseline data for treatment and placebo per cycle will be determined. The means and 95% confidence intervals (CIs) for the differences will be calculated within treatment pairs for each outcome. The N-of-1 trials will be combined using a hierarchical Bayesian effects model to estimate the average effect that incorporate variance within- and between-individuals.

Sample size. A sample size of 8 participants will provide a power of 80% to detect a minimal clinically important difference (MCID) of change in CRP (≥ 35% reductions in this trial). A maximum of 10 participants will be enrolled (dropout rate of 20%). The estimation was based on the Yang et al. equations and implemented into an R Shiny app [https://jiabeiyang.shinyapps.io/SampleSizeNof1/].

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset cancer survivors with a diagnosis of breast, colon, colorectum, rectum, prostate, non-small lung, Hodgkin lymphoma, non-Hodgkin lymphoma, chronic lymphoid leukaemia and chronic myeloid leukaemia cancer.
* Aged ≥ 18 years at cancer diagnosis -upper age limit to study entry = 75 years.
* People of both genders, all racial and ethnic backgrounds.
* Non-smokers (i.e., not smoking during previous 12 months).
* A history of local, regional or distant recurrence, primary second cancers or multiple primary tumours will be not reasons to exclude.
* No previous evidence for metastatic disease.
* Evidence of complete remission defined as a decrease in or disappearance of signs and symptoms of cancer after treatment.
* Having completed definitive treatment (surgery, neoadjuvant/adjuvant cytotoxic chemotherapy, radiotherapy, immunotherapy) at least 12 months.
* Continuous, maintenance therapy is considered if initiated ≥3 months prior to study treatment and prescribed for long-term, chronic use without interruption during the trial, or completed for at least ≥3 months before starting the trial.
* Having a high inflammatory cardiac risk profile at the initial screening defined as a CRP measurement ≥ 3 to < 10 mg/L, or ≥ 10 mg/L if acute inflammation is ruled out.
* Having stable hypertension (if applicable): no medication changes in prior 30 days, systolic BP <160 mm Hg and either ≥ 130 mm Hg without antihypertensive medications, or diagnosis of hypertension in medical records.
* Clinical evidence of cardiovascular, respiratory and/or musculoskeletal disease, and/or other controlled and stable chronic medical conditions will not be reason of exclusion.
* Any medical prescription(s) if routinely administered and continued through the trial period.
* Living at one of the urban areas of the city of Valencia with the highest index impact of pollutant on population values (IIPP > 125): Russafa, Malilla and Arrancapins neighbourhoods.
* Permanent residence in their usual home at least 3 months prior to the first collected blood sample in the first cycle and without plans to move out toward another dwelling during the trial study.
* Living in a non-smoking household.
* Internet connection (Wi-Fi) in the house.
* Signed informed consent prior to commencement of specific protocol procedures.

Exclusion Criteria:

* Recently diagnosed with cancer or plans for additional cancer therapy and/or surgery during the trial period.
* Metastatic disease.
* Planned medication prescription to start during the trial.
* Current chronic anti-inflammatory drug prescriptions or other chronic drugs (e.g., antihypertensive drugs) will be no reason for exclusion if its use is continued for the duration of the trial period.
* Having uncontrolled hypertension: participants with average systolic BP >160 mmHg over any 10-day period prior and during the study.
* History of uncontrolled, unstable chronic disease as defined by clinical practice guidelines and documented in medical records - within past 6 months to screening visit(s) and during the study (i.e., uncontrolled diabetes mellitus). Psychiatric illness that would limit compliance with trial requirements and/or prevent the patient from giving informed consent.
* History of ongoing, chronic or recurrent infectious disease, and having suspected or proven immunocompromised state (i.e., Human Immunodeficiency Virus infection).
* Self-report of alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of more than 14 alcoholic drinks per week).
* Shift workers or subjects who have the work schedule falling outside the hours of 07:00 a.m. and 10:00 p.m.
* Plans to move out of usual home during the trial period.
* Unwilling to spend at least 7-h/overnight in the bedroom.
* Pre-existing an air filtration system that improve household air quality. If so, the device will be disconnected during all the trial cycles.
* Unwilling to give consent.

Additional inclusion criteria (non-exclusive; when CRP test is unavailable in medical records) associated with high or very high cardiovascular (CV) toxicity risk factors (according to the European Society of Cardiology guidelines on Cardio-Oncology):

1. High or very high baseline CV toxicity risk pre-treatment (HFA-ICOS risk stratification score); risk factors including:

   * Prior history of CV disease (e.g., coronary artery disease).
   * Presence of multiple CV-risk factors (e.g., hypertension, dyslipidemia).
   * Current or concomitant cancer treatment.
   * Prior cardiotoxic cancer therapy (e.g., anthracycline, radiotherapy to left chest).
   * Lifestyle risk factors (history of smoking, body mass index >30).
2. Specific cardiotoxic cancer therapies with a high risk of long-term CV complications (any of these):

   * Total lifetime cumulative dose anthracycline ≥ 250 mg/m2 doxorubicin equivalent.
   * High-dose anthracycline ≥ 250 mg/m2 doxorubicin equivalent.
   * High-dose RT > 15 Gray (Gy) Mean Heart Dose (MHD).
   * Anthracycline ≥ 100 mg/m2 doxorubicin equivalent in combination with radiotherapy 5-15 Gy MHD.
   * Multitargeted tyrosine kinase inhibitors (TKI) targeting BCR-ABL and concomitant high-dose dexamethasone therapy >160 mg/month.
   * Combination of RAF and MEK inhibition.
   * Single-agent immune checkpoints inhibitors (ICI) therapy followed by previous cardiotoxic cancer therapies: RT, anthracyclines, 5-fluorouracil, and TKI.
   * Combination of two types of ICI (anti-PD1, e.g., nivolumab and anti-CTLA-4, e.g., ipilimumab).
3. Moderate or severe cancer therapy-related CV toxicity detected during cancer treatment or new CV symptomatic/asymptomatic abnormalities at the end of cancer treatment (3 or 12 months after therapy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein (CRP) | At baseline and in the day 7 and 14 of each period. In the same time interval in the morning (between 07:00-10:00 am).
  The primary outcome is the change in blood CRP concentrations. A portable point-of-care testing via capillary finger-prick microsampling will be used to measure the blood levels of CRP (5µl per participant once a week; measuring range, 0.48-200 mg/L).

SECONDARY OUTCOMES:
D-dimer | At baseline and in the day 7 and 14 of each period. In the same time interval in the morning (between 07:00-10:00 am).
  Changes in the blood levels of D-dimer. A portable point-of-care testing via capillary finger-prick microsampling will be used to measure the blood levels of D-dimer (30µl per participant once a week; measuring range, 0.1-10 µg/mL).
Serum Amyloid A (SAA) | At baseline and in the day 7 and 14 of each period. In the same time interval in the morning (between 07:00-10:00 am).
  Changes in the blood levels of SAA. A portable point-of-care testing via capillary finger-prick microsampling will be used to measure the blood levels of SAA (5µl per participant once a week; measuring range, 2-300 µg/mL).
Haemoglobin A1c (Hb1Ac) | At baseline and in the day 7 and 14 of each period. In the same time interval in the morning (between 07:00-10:00 am).
  Changes in the blood levels of Hb1Ac. A portable point-of-care testing via capillary finger-prick microsampling will be used to measure the blood levels of Hb1Ac (5µl per participant once a week; measuring range, 3%-14%).
Systolic and diastolic blood pressure (BP) | At baseline and in the day 7 and 14 of each period. In the same time interval in the morning (between 07:00-10:00 am) and before the blood collection and any medication and in a fasting condition.
  Changes in the peripheral systolic and diastolic BP . Self-measurements of BP will be taken by the participants using a portable upper-arm cuff oscillometric device. The mean of 3 automated BP readings taken at 60-sec intervals will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Mallilla Primary Care Practice, Valencia
  - Russafa Primary Care Practice, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Identifiable information will not be shared with any partners, either during, or after the completing of the trial. However, anonymous data will be made accessible by the study collaborators based inside the UK and outside the European Economic Area, and for research analysis purposes and revision of manuscripts to publication(s). Research datasets will be pseudonymised by using a random ID code number assigned to each participant and keeping separately the data and the identifiers. Only the pseudonymised data will be shared with the study collaborators, and thus, they will only work with anonymised project files. These will be uploaded into the REDCap project's File Repository and sent securely via UCL REDCap Services using its Send-It application. File download is performed over an SSL encrypted connection.
  The database system used for this research project will be created using UCL REDCap Services.
Supporting Information: Study Protocol
Access Criteria: Access to all information systems will be controlled to ensure that only authorised users have access to the system and the information they are authorised to access. Only the Field Researcher (Eva Hernandez-Garcia) and Principal Investigator (Emeritus Professor Andrew Edkins) will have complete access to the database.